CLINICAL TRIAL: NCT01544335
Title: Evaluation of the Validity of BIS as a Tool for Quantification of Lymphedema Through Comparison With Perometry and Self-Report
Brief Title: Evaluation of BIS for Quantification of Lymphedema
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alphonse Taghian, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 11-325
Record Dates: First submitted 2012-02-12; First posted 2012-03-05 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- BIS: Subjects evaluated using Bioimpedance Spectroscopy
  Interventions: Other: Bioimpedance Spectroscopy

INTERVENTIONS:
Other: Bioimpedance Spectroscopy — BIS used to measure fluid in arm

SUMMARY:
The purpose of this study is to determine whether measuring the fluid in your arms using Bioimpedance Spectroscopy is as effective at detecting and monitoring lymphedema as measurements with the Perometer. The investigators will also evaluate any symptoms you may experience in your arms during and after treatment for breast cancer with a questionnaire.

DETAILED DESCRIPTION:
During the study whenever you have an arm volume measurement using the Perometer, we will also measure the fluid in your arms using Bioimpedance Spectroscopy. These measurements are made by passing a harmless electrical signal of very low strength through your body to determine the difference in the amount of fluid in each arm. The test is simple and painless, and takes about 3 minutes. In addition, whenever you have an arm measurement, you will be asked to complete a questionnaire. While completing the questionnaire, you can skip any questions you do not wish to answer. The questionnaires will take about 10 minutes to complete. Arm measurements with the Perometer and Bioimpedance Spectroscopy and completion of the questionnaire will occur every 4-7 months when you are at MGH for regular medical visits.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive or in-situ carcinoma of the breast
* Participants must have undergone sentinel node mapping or axillary dissection
* Life expectancy of greater than 1 year.
* Willingness to comply with required follow up Perometer and BIS measurements and completion of LEFT-BC questionnaire

Exclusion Criteria:

* Patients who have known metastatic disease or other locally advanced disease in the thoracic or cervical regions
* Any patient who will not be returning routinely for follow-up at MGH or DFHCC
* Participants with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of primary lymphedema
* History of prior surgery or radiation to the head, neck, upper limb, or trunk
* Participants who have evidence that axillary lymph node malignancy is causing lymphedema due to recurrence as per physician discretion
* Any patient who has bilateral lymph node mapping or dissection
* Any patient with a current case of cellulitis
* Patients with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with histologically or cytologically confirmed breast cancer who will be returning routinely for follow-up at Massachusetts General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2011-12; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Gillespie TC, Roberts SA, Brunelle CL, Bucci LK, Bernstein MC, Daniell KM, Naoum GN, Miller CL, Taghian AG. Comparison of perometry-based volumetric arm measurements and bioimpedance spectroscopy for early identification of lymphedema in a prospectively-screened cohort of breast cancer patients. Lymphology. 2021;54(1):1-11. PMID 34506083
- See also: Gillespie 2021 Publication Link — https://pubmed.ncbi.nlm.nih.gov/34506083/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 270 participants were accrued, however 65 had to be excluded because they later received bilateral breast surgery and 14 withdrew consent. This is why 191 participants started the study.
Groups:
- Bioimpedance Sprectroscopy: Subjects evaluated using Bioimpedance Spectroscopy
  Bioimpedance Spectroscopy: BIS used to measure fluid in arm
Period: Overall Study
Arm/Group | Bioimpedance Sprectroscopy
Started | 191
Completed | 138
Not Completed | 53
Not completed — Lost to Follow-up | 27
Not completed — Death | 4
Not completed — Disease progression | 3
Not completed — Baseline Measurements not Available | 19

BASELINE CHARACTERISTICS:
Population: Participants included in analysis who had at least one post-operative follow up measurement
Groups:
- Bioimpedance Spectroscopy: Subjects evaluated using Bioimpedance Spectroscopy
  Bioimpedance Spectroscopy: BIS used to measure fluid in arm
Arm/Group | Bioimpedance Spectroscopy
Number analyzed (Participants) | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 111
  >=65 years | 27
Age, Continuous [Median (Full Range); unit: years] | 53.7 [27.2 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 138

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Impedance Ratios Obtained Through Bioimpedance Spectroscopy (BIS) With Perometric Relative Arm Volume Change (RVC)
Description: Correlation of volumetric measurements obtained using Perometry with impedance ratios obtained through BIS at the baseline examination and during follow-up visits. Impedance ratios will also be correlated with symptoms indicated in the LEFT-BC questionnaires completed during each examination. Volumetric arm measurements from perometry will be quantified using the RVC formula, which will be compared with impedance ratios calculated using the BIS device software.
Time Frame: 5 years
Population: 53 of the 191 participants had to be excluded. 27 lost to follow up, 4 died on the study, 3 had disease progression, and baseline measurements were not available for 19 participants.
Measure: Number; unit: correlation coefficient
Units Other Than Participants: measurements
Arm/Group | Bioimpedance Sprectroscopy
Number analyzed (Participants) | 138
Number analyzed (measurements) | 442
correlation coefficient | 0.195
Statistical Analysis 1: Comparison: Bioimpedance Sprectroscopy; Test type: Other; p < 0.001, Correlation coefficient; The correlation between RVC and ΔL-Dex values was plotted, and the correlation strength was assessed using the Pearson correlation coefficient, r

2. Secondary Outcome: Compare Relationship Between Lymphedema Diagnostic Criteria Corresponding to BIS, Perometry, and Self-reported Symptoms
Description: Relationship among diagnostic criteria pertaining to BIS, perometry, and self-reported symptoms. A change of >3 Standard Deviations in impedance ratios compared to pre-surgical baseline is considered diagnostic for lymphedema when BIS is utilized. A relative volume change of >5% - >10% compared to baseline is considered lymphedema by perometry. Self-report of symptoms including feelings of swelling, heaviness, and tightness are often considered as criteria for lymphedema.
Time Frame: 5 years
Population: This data was not collected and outcome cannot be reported.
Arm/Group | Bioimpedance Sprectroscopy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Bioimpedance Spectroscopy
All-Cause Mortality (participants affected / at risk) | 4/191
Serious Adverse Events (participants affected / at risk) | 0/191
Other Adverse Events (participants affected / at risk) | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT01544335/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT01544335/ICF_001.pdf